CLINICAL TRIAL: NCT01552369
Title: Prophylaxis Versus Preemptive Therapy for the Prevention of CMV in High-Risk R-D+ Liver Transplant Recipients
Brief Title: CMV Antiviral Prevention Strategies in D+R-Liver Transplants ("CAPSIL")
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0073
Record Dates: First submitted 2012-03-02; First posted 2012-03-13 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2018-03-22

CONDITIONS: Cytomegalovirus Infection
Keywords: CMV; cytomegalovirus infections; ganciclovir; liver transplant; preemptive therapy; prophylaxis; valganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Valganciclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preemptive Therapy (Experimental): 900 mg of Valganciclovir given orally twice daily to Preemptive Therapy subjects upon detection of CMV viremia until plasma PCR is negative on two consecutive weekly PCR test. All dosages adjusted for renal dysfunction. n=88
  Interventions: Drug: Valganciclovir
- Prophylaxis (Active Comparator): 900 mg of Valganciclovir given orally once daily to subjects for 100 days post transplantation. All dosages adjusted for renal dysfunction. n=88
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir, 900 mg given orally once daily to all Prophylaxis group subjects for 100 days post transplantation as prophylaxis. Valganciclovir, 900 mg given orally twice daily to Preemptive Therapy group subjects as a PET only after a positive CMV PCR test and stopped after PCR is negative for 2 consecutive weeks.

SUMMARY:
This is a trial of preemptive therapy vs. prophylaxis for prevention of Cytomegalovirus (CMV) disease in R-D+ liver transplant patients. Subjects will be randomized within 10 days of transplant to receive in an open label design, either antiviral prophylaxis with valganciclovir, 900 mg orally once daily or preemptive therapy (weekly monitoring for CMV viremia by plasma PCR) for 100 days post-randomization with initiation of oral valganciclovir 900mg orally twice daily at onset of CMV viremia and continued until plasma PCR is negative on two consecutive weekly PCR tests). A minimum of 176 subjects will be enrolled in the study. The study duration is 7 years. The primary objective of this study is to compare prophylaxis versus preemptive therapy using valganciclovir for the prevention of CMV disease in R-/D+ liver transplant recipients.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter trial of preemptive therapy vs. prophylaxis for prevention of Cytomegalovirus (CMV) disease in seronegative recipient- seropositive donor (R-D+) liver transplant patients.Subjects will be randomized within 10 days of transplant to receive in an open label design, either antiviral prophylaxis with valganciclovir 900 mg orally once daily or preemptive therapy for 100 days post-randomization with initiation of oral valganciclovir 900mg orally twice daily at onset of CMV viremia (monitored weekly) and continued until plasma PCR is negative on two consecutive weekly PCR tests. Study participants will be followed during the intervention period (100 days post randomization) and until 12 months post-transplant for CMV disease, toxicity, and clinical outcomes (opportunistic infections, rejection, graft loss and mortality). Drug safety labs will be assessed and recorded for the entire treatment period in both the prophylaxis and preemptive group. Re-transplantation and all-cause mortality will also be assessed at study closure and no longer than 5 years after enrollment. Additionally, the impact of the two CMV prevention strategies on CMV-specific cellular and humoral immune responses will be evaluated at 100 days after randomization, and 6 and 12 months post-transplant. A minimum of 176 subjects will be enrolled in the study. Allowing for over-enrollment to replace dropouts, up to 205 subjects may be enrolled to achieve the target enrollment of 176. Subjects will be randomized into one of the two groups in 1:1 ratio. The study duration is 7 years. The primary objective of this study is to compare prophylaxis versus preemptive therapy using valganciclovir for the prevention of CMV disease in R-/D+ liver transplant recipients. The secondary objectives are:1) to assess the two preventive strategies for clinical outcomes (major bacterial, fungal and non-CMV viral infections, rejection, graft loss and mortality) at one year post transplantation; 2) to assess the two preventive strategies for hematologic toxicity (assessment of neutropenia and receipt of hematopoietic growth factor during study days 1-107).

ELIGIBILITY:
Inclusion Criteria:

1. Be > / = 18 years of age.
2. Have negative Cytomegalovirus (CMV) serology (confirmed within 6 months of transplant) and receive a liver from a donor with positive CMV serology (R-/D+).
3. Have received their first orthotopic liver transplant (the transplanted liver may be deceased donor or live donor graft) within 10 days prior.
4. Have absolute neutrophil count > 1000/µL at randomization.
5. - If female, and not postmenopausal or surgically sterile, must have negative pregnancy test (serum or urine) within 48 hours prior to randomization and must also agree to use medically approved method of contraception. Acceptable methods include: barrier method, intrauterine device (hormonal or non-hormonal), oral hormonal contraceptives, abstinence for 100 days after randomization and 3 months after valganciclovir cessation.

   -- If male, and has not had a vasectomy, he must agree to practice barrier method of contraception for 100 days after randomization and 3 months after valganciclovir cessation.
6. Subject or legally authorized representative has provided written informed consent.

Exclusion Criteria:

1. Currently enrolled in any interventional trial of an investigational therapeutic agent unless co-enrollment has been approved by study Principal Investigators (PIs) and the DMID prior to enrollment.
2. Have hypersensitivity to acyclovir, ganciclovir or valganciclovir.
3. Be breast-feeding mother.
4. Have known Human immunodeficiency virus (HIV) infection (based on testing performed during the transplant evaluation process).
5. Be undergoing multi organ transplant or have undergone prior organ transplant.
6. Have expected life expectancy of less than 72 hours.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - Emory Clinic - Transplant Center, Atlanta, Georgia
  - Mayo Clinic, Rochester - Infectious Diseases, Rochester, Minnesota
  - Mount Sinai School of Medicine - Medicine - Infectious Diseases, New York, New York
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - University of Washington - Medicine, Seattle, Washington

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Singh N, Winston DJ, Razonable RR, Lyon GM, Silveira FP, Wagener MM, Limaye AP. Risk Factors for Cytomegalovirus Viremia following Liver Transplantation With a Seropositive Donor and Seronegative Recipient Receiving Antiviral Therapy. J Infect Dis. 2021 Mar 29;223(6):1073-1077. doi: 10.1093/infdis/jiaa470. PMID 32726431
- [Derived] Singh N, Winston DJ, Razonable RR, Lyon GM, Silveira FP, Wagener MM, Stevens-Ayers T, Edmison B, Boeckh M, Limaye AP. Effect of Preemptive Therapy vs Antiviral Prophylaxis on Cytomegalovirus Disease in Seronegative Liver Transplant Recipients With Seropositive Donors: A Randomized Clinical Trial. JAMA. 2020 Apr 14;323(14):1378-1387. doi: 10.1001/jama.2020.3138. PMID 32286644

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 538 liver transplant candidates or recipients were screened. 333 were not eligible. 229 did not meet inclusion criteria. 29 met at least 1 exclusion criteria. 75 unable to give, or refused consent. No study procedures were conducted on these 333 subjects.
Groups:
- Preemptive Therapy: 900 mg of Valganciclovir given orally twice daily to Preemptive Therapy subjects upon detection of CMV viremia until plasma PCR is negative on two consecutive weekly PCR test. All dosages adjusted for renal dysfunction. n=100
- Prophylaxis: 900 mg of Valganciclovir given orally once daily to subjects for 100 days post transplantation. All dosages adjusted for renal dysfunction. n=105
Period: Overall Study
Arm/Group | Preemptive Therapy | Prophylaxis
Started | 100 | 105
One Year (Subjects completed major endpoints; CMV disease and/or all-cause mortality) | 100 | 105
Final Follow up | 92 | 96
Completed (Subjects that completed major endpoint; CMV disease and/or all-cause mortality) | 92 | 96
Not Completed | 8 | 9
Not completed — Did not consent to extended follow up | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preemptive Therapy | Prophylaxis | Total
Number analyzed (Participants) | 100 | 105 | 205
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [49.5 to 62.5] | 58 [51 to 63] | 58 [50 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 27 | 62
  Male | 65 | 78 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 92 | 94 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 90 | 99 | 189
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 100 | 105 | 205
Baseline absolute neutrophil count(ANC) [Mean (Inter-Quartile Range); unit: Count per 1000 cells/µL] — ANC collected prior to the initiation of intervention
  Count per 1000 cells/µL | 6888 [3500 to 8640] | 7409 [3600 to 9640] | 7160 [3600 to 9325]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Cytomegalovirus (CMV) Disease.
Description: CMV disease as verified by an independent end point committee
Time Frame: 365 days post-transplant
Population: All randomized subjects
Measure: Number; unit: participants
Groups:
- Preemptive Therapy: 900 mg of Valganciclovir given orally twice daily to Preemptive Therapy subjects upon detection of CMV viremia until plasma PCR is negative on two consecutive weekly PCR test. All dosages adjusted for renal dysfunction.
- Prophylaxis: 900 mg of Valganciclovir given orally once daily to subjects for 100 days post transplantation. All dosages adjusted for renal dysfunction.
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
participants | 9 | 20
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.0396, Mantel Haenszel
Statistical Analysis 2: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.048, Competing risk regression; Death was considered a competing risk; Hazard Ratio (HR) = 2.22, 95% CI 2-sided [1.01 to 7.3] — The risk of CMV disease is 2.2x higher in the prophylaxis group when compared to the preemptive group

2. Secondary Outcome: All-cause Mortality
Description: Survival probability at 1 year
Time Frame: Up to 365 days post-transplant
Population: Intent to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: survivor probabillity
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
survivor probabillity | .880 [.798 to .930] | .933 [.865 to .967]
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority — log-rank test for equality of survivor functions; p = 0.19, Log Rank

3. Secondary Outcome: Incidence of Allograft Rejection
Description: Number of subjects with allograft rejection
Time Frame: Up to 365 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 28 | 26
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.60, Mantel Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.45 to 1.58] — The odds of rejection in prophylaxis group compared to preemptive group

4. Secondary Outcome: Graft Loss
Description: Incidence of graft loss (re-transplantation)
Time Frame: Up to 365 days post-transplant
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 2 | 2
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.96, Mantel Haenszel; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.13 to 6.92] — The odds of graft loss in prophylaxis group compared to preemptive group

5. Secondary Outcome: Late-onset CMV Disease
Description: Incidence of late-onset CMV disease (occurring after 100 days post-randomization) as adjudicated by end point committee
Time Frame: Up to 365 days post-transplant
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 6 | 18
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.014, Mantel Haenszel; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.21 to 8.69] — Odds of late disease in prophylaxis group compared to preemptive

6. Secondary Outcome: Bacterial Infections
Description: Incidence of bacterial opportunistic infections
Time Frame: Up to 365 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 22 | 26
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.64, Mantel Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.61 to 2.23] — Odds of bacterial infection in prophylaxis subjects compared to preemptive

7. Secondary Outcome: Major Fungal Infections
Description: Opportunistic fungal infections
Time Frame: Up to 365 days post-transplant
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 4 | 9
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.18, Mantel Haenszel; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.66 to 7.62] — Odds of fungal disease in prophylaxis group compared to preemptive

8. Secondary Outcome: Major Non-CMV Viral Infections
Description: Incidence of non-CMV viral infections
Time Frame: Up to 365 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 2 | 0
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.24, Fisher Exact

9. Secondary Outcome: Neutropenia
Description: Incidence of neutropenia less than 1000/µL while on valganciclovir treatment
Time Frame: Day 1 through Day 107
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 36 | 35
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.69, Chi-squared

10. Secondary Outcome: Neutropenia Less Than 500
Description: ANC less than 500 while on valganciclovir
Time Frame: prior to day 107
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 12 | 10
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.57, Chi-squared

11. Secondary Outcome: Hematopoietic Growth Factors
Description: Hematopoietic growth factor receipt for ANC less than 500 during valganciclovir treatment.
Time Frame: Day 1 through Day 107
Measure: Count of Participants; unit: Participants
Arm/Group | Preemptive Therapy | Prophylaxis
Number analyzed (Participants) | 100 | 105
Participants | 5 | 7
Statistical Analysis 1: Comparison: Preemptive Therapy vs Prophylaxis; Test type: Superiority; p = 0.61, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Description: Liver transplant recipients represent a population in whom a high rate of medical events are commonly seen during the post-transplant course. For this study, adverse events were:
  Any clinically important untoward medical occurrence in a subject receiving study drug that is different from what is expected in the clinical course of a patient with a liver transplant.
  Any clinically important, untoward medical occurrence thought to be related to the study drug, regardless of 'expectedness'.
Arm/Group | Preemptive Therapy | Prophylaxis
All-Cause Mortality (participants affected / at risk) | 12/100 | 7/105
Serious Adverse Events (participants affected / at risk) | 2/100 | 0/105
Other Adverse Events (participants affected / at risk) | 1/100 | 1/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preemptive Therapy (N=100) | Prophylaxis (N=105)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preemptive Therapy (N=100) | Prophylaxis (N=105)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT01552369/Prot_SAP_000.pdf